CLINICAL TRIAL: NCT03382444
Title: A Longitudinal Assessment of Cognitive Impairment in Advanced CKD Transitioning Into Renal Replacement Therapy
Brief Title: The Kidney and The Brain Study - Assessment of Cognitive Impairment in Advanced CKD
Status: Completed | Type: Observational
Sponsor: Natalie Garratt (Other)
Responsible Party: Sponsor-Investigator, Natalie Garratt, Research Development Lead, Northern Care Alliance NHS Foundation Trust
Organization: Northern Care Alliance NHS Foundation Trust (Other)
Other Study IDs: 17/233064-S
Record Dates: First submitted 2017-09-29; First posted 2017-12-26 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Cognitive Impairment; Chronic Kidney Diseases; End Stage Renal Disease; Dementia; Hemodialysis Complication; Peritoneal Dialysis Complication; Renal Transplant
Keywords: cognitive impairment; hemodialysis; dementia; end stage renal disease
MeSH Terms: conditions — Cognitive Dysfunction; Renal Insufficiency, Chronic; Kidney Failure, Chronic; Dementia | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cognitive Assessment — Each patient with have a 2 hour cognitive assessment at baseline, 3months after starting renal replacement therapy and 12 months after starting renal replacement therapy
Diagnostic Test: Depression and Quality of Life Assessment — Each patient with have a 2 hour depression and QOL assessment at baseline, 3months after starting renal replacement therapy and 12 months after starting renal replacement therpay

SUMMARY:
Patients with failed kidneys need Renal Replacement Therapy (RRT) to remove fluid and toxins from the body. The 3 types of RRT are kidney transplant or removal of waste by dialysis, either via the blood (haemodialysis) or via the stomach area (peritoneal dialysis). 27,000 patients currently receive dialysis in the UK and some endure reduced quality-of-life, depression, and thinking and memory difficulties. Some of these symptoms reflect undiagnosed dementia. Indeed up to 7/10 dialysis patients suffer moderate to severe brain impairment or dementia - much more frequently than in the general population.

This study will assess brain function just before starting dialysis/transplant and at 3 and 12 months afterwards with face to face assessments and with brain scans in some patients. Changes in brain function will be compared between people treated with the different forms of dialysis and transplant.

The Investigators hope to evaluate whether these tests are acceptable to patients, whether affected sub-groups with cognitive impairment can be identified early, and if certain dialysis methods are better for patients with cognitive impairment/dementia, so that a larger study to try to improve brain function after RRT can be developed.

DETAILED DESCRIPTION:
Aims of the proposed research

Primary Objective:

To test the feasibility of performing serial detailed neurocognitive assessments in patients before during and after the period of commencing RRT for End-Stage Kidney Disease

Secondary Objectives:

1. Estimate cross-sectional and longitudinal variability in a novel battery of neurocognitive assessments amongst participants in transition to all 3 modalities of RRT.
2. Assess the administration, suitability and adherence of the chosen cognitive and quality of life measures in participants.
3. Test the feasibility of recruitment to a longitudinal brain magnetic resonance imaging (MRI) study in a randomly selected proportion of participants.
4. Estimate the cross-sectional and longitudinal variability in multiparametric brain MRI parameters and their interaction with cognitive functional change in this transitional population.
5. To describe resource implications including patients referred to specialist services due to new diagnoses of cognitive impairment, dementia and/or depression

Study Design

This is a prospective study of 96 patients who are about to commence renal replacement therapy (RRT). Patients will undergo a neurocognitive, depression and quality of life assessments at baseline, 3 months after commencing RRT and 12 months after commencing RRT. A nested cohort of 25% will undergo MR brain scans at baseline and at 12 months.

Detailed Plan of Investigation

Recruitment procedure The target population is clinic based patients with advanced CKD who are due to commence RRT in the next 1-2 months as determined by the treating clinician. Patient screening, information giving and consenting for this feasibility study will be performed in the low clearance clinic at Salford (held twice per week). Enrolment of willing and eligible patients who are admitted into hospital to start RRT in the absence of infection and delirium may also be assessed.

Study Protocol Overall feasibility of the study will be assessed based on recruitment rates of eligible patients as well as consent rates, withdrawal rates, missing data and study costs. This data is also relevant to assess the feasibility of performing brain MR scans in this cohort. In addition, factors which may impact on cognitive function, such as age, gender, education, ethnicity and socioeconomic status, will be assessed at baseline to better inform future trial design.

Participants will undergo testing of all measures (except imaging) at baseline, 3 months after starting renal replacement therapy (RRT+3) and after 12 months (RRT+12). Baseline is defined as any participant whose eGFR is <15mls/min/1.73m2 and is expected to need to start renal replacement therapy within 2 months. An opportunistic sampling technique will be used. The research fellow will engage in multidisciplinary meetings that follow the low clearance clinics and will use these to identify potential participants, participants will then be contacted and if they demonstrate potential willingness to participate then will be sent the participant information sheet. Consent will then be taken and if the participant is expected to start RRT within 2 months then baseline assessments will occur at next clinic appointment.

Where participants transfer from one modality of dialysis to another the participants will be assigned to the modality of dialysis most frequently undertaken in the 3 months prior to testing. Assessment will be delayed when there has been a modality switch within the last 1 month of assessment date. Where a participant has received a renal transplant after commencing dialysis cognitive assessment will occur as near to the 3 and 12-month time point as possible. Where a participant receives a pre-emptive transplant (prior to any dialysis) then cognitive assessments will occur at 3 and 12 months post-transplant date.

Cognition Cognitive assessments will be performed by the research fellow in a quiet clinical room with refreshments made available to the participants. This methodology has been used previously. Family members or carers will not be present. The assessments may last up to 2 hours. The assessments will usually follow clinic appointments to minimise participant inconvenience. Due to fluctuations in cognition in the weekly haemodialysis cycle. Cognitive assessments will occur on non-dialysis days in participants undergoing haemodialysis. There are no known treatment related fluctuations in cognition in peritoneal dialysis and these participants will be assessed before or after routine clinic appointments. The neurocognitive tests will be a combination of previously used and validated tests (below) and specifically designed assessments by Professor Montaldi at University of Manchester. They will be designed to detect the expected defects in cognitive domains that are known to be present in CKD and dialysis patients. It will be probe into these defects with more thoroughness and sensitivity than has been undertaken in previous studies.

The MoCA is a one-page 30-point screening test of global cognitive function taking approximately 10 minutes to administer. There are 3 alternate forms in English designed to minimize practice effects in longitudinal studies. The MoCA will be used in this study primarily to allow comparison with the results of other studies in RRT. It will also permit the first longitudinal validation of the MoCA in the target group against our detailed neurocognitive battery.

The main standardised neurocognitive tests will include:

* IQ (WASI);
* Memory (Weschler Memory Scale, Doors and People, Rey Figure) subtests;
* Speed of processing, attention (TEA) and executive function subtests (Hayling and Brixton).

Detection of more subtle memory changes over time will be explored using a similar foils test designed by Montaldi and colleagues and used in an older population The neurocognitive battery will be especially optimised to avoid potential practice effects.

Anxiety and Depression There are complex interactions between anxiety, depression and cognition. This has also been demonstrated in a cohort of haemodialysis patients. The hospital anxiety and depression scale will be used to measure this confounding variable. It has been used in a similar fashion in other studies of similar patient populations. It takes the form of a questionnaire and takes 2-5 minutes to complete. A systematic review of this tool identified that a score of 8/21 was optimal for the balancing sensitivity and specificity of an accurate depression and anxiety diagnosis. Participants with newly diagnosed severe anxiety or depression will be referred onwards to our renal psychology teams and local mental health care providers as appropriate.

Quality of life Quality of life (QOL) is an important output of healthcare analyses with quality of life factoring into patient decisions on RRT modality choices. A meta analyses of healthcare related quality of life demonstrated that in-centre haemodialysis patients suffered most. However most studies are cross sectional and subject to ascertainment bias. This study will use KDQOL-36TM questionnaire. This is a purposely designed QOL instrument for patients on dialysis. Relevant questions will be used at month 0 and the whole instrument will be applied at month RRT+3 and RRT+12.

Magnetic Resonance brain imaging Clinicians need to identify which patients are susceptible to cognitive changes in the future. Similarly, our renal service user group identified dementia risk as a key patient concern. Neuroimaging at baseline will identify those with changes indicative of vulnerability to cognitive decline. Longitudinal MR changes will provide insight into mechanistic aetiology and will help clarify the link between brain structure and function.

The Investigators will use a state-of the art dementia imaging protocol in a randomly selected group of 25% participants. This protocol has been developed by Dr Parkes and others as part of the Dementia Platforms UK Imaging network. This includes measures of gross morphological structure from high resolution T1-weighted images, microstructural change from diffusion-weighted imaging and markers of microvascular disease from T2-weighted FLAIR imaging (to quantify white matter lesion volume), susceptibility-weighted imaging (to visualise microbleeds) and arterial spin labelling (ASL) (for cerebral blood flow images). These quantitative imaging measurements will provide insight into the mechanisms by which kidney disease impacts cognition, and may allow prediction of the progression of such impairment. In particular, ASL (a technique in which Dr Parkes is internationally renowned), will provide information on the metabolic state of the brain which may be altered in kidney disease. Advanced diffusion-weighted imaging will also provide a sensitive indicator of loss of neural density/structure. The imaging protocol will last for 45 minutes and studies will be carried out in the MR imaging facilities at Central Manchester University Hospital, using exactly the same protocol. MR imaging will be performed twice in each of these participants - first prior to commencement of RRT and within 1 month of the baseline cognitive assessment and then within1 month of the RRT +12 assessment

ELIGIBILITY:
Inclusion Criteria:

1. eGFR <15/ml/min/1.73m2
2. Aged 55 years and over
3. Mental capacity to understand the study and give informed consent

Exclusion Criteria:

1. Age <55 years
2. Non-English speaking
3. Patients known to have a psychiatric condition, including severe depression, bipolar affective disorder, severe anxiety, panic disorder, substance misuse or psychosis or previous severe head injury
4. Contraindications to magnetic resonance imaging
5. Patients who have chosen not to undergo dialysis treatment (conservative care).

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is clinic based patients with advanced CKD who are due to commence RRT in the next 1-2 months as determined by the treating clinician. Patient screening, information giving and consenting for this feasibility study will be performed in the low clearance clinic at Salford (held twice per week). Enrolment of willing and eligible patients who are admitted into hospital to start RRT in the absence of infection and delirium may also be assessed.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
To test the feasibility of performing serial detailed neurocognitive assessments in patients before during and after the period of commencing RRT for End-Stage Kidney Disease | 2.5years
  Number of patients eligible, no of patients consented, number of patients who underwent both baseline and longitudinal neurocognitive assessments

SECONDARY OUTCOMES:
Estimate cross-sectional and longitudinal variability in a novel battery of neurocognitive assessments amongst participants in transition to all 3 modalities of RRT. | 2.5years
  Determine variability in global cognitive scores and domain specific scores at baseline and then longitudinal trajectories at RRT+3months and RRT+12months
Assess the administration, suitability and adherence of the chosen cognitive and quality of life measures in participants. | 2.5 years
  Number of patients who agree to undertake all cognitive assessments, quality of life assessments and depression assessments as a total of the number of patients who participate
Test the feasibility of recruitment to a longitudinal brain magnetic resonance imaging (MRI) study in a randomly selected proportion of participants. | 18 months
  Number of patients who undergo MR brain scans at baseline and at RRT+12months as a proportion of patients eligible and patients who undergo cognitive assessment.
Estimate the cross-sectional and longitudinal variability in multiparametric brain MRI parameters and their interaction with cognitive functional change in this transitional population. | 2.5years
  Quantitative imaging maps of microstructure (from diffusion-weighted images) and cerebral blood flow will be co-registered to the T1-weighted image and median values extracted from each region of interest, along with volumes from the T1-weighted image. In addition, the number of microbleeds and the white matter lesion volume will be recorded.
To describe resource implications including patients referred to specialist services due to new diagnoses of cognitive impairment, dementia and/or depression | 2,5 years
  To record the number of patients who are referred for specialist assessment for their cognitive impairment and/or depression

CONTACTS AND LOCATIONS:
Overall Officials: James Tollitt, MBcHB, Principal Investigator — Northern Care Alliance NHS Foundation Trust
Locations (1):
- Salford Royal Nhs Foundation Trust, Salford, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No